# Statistical Analysis Plan

March 20, 2023

**Title** Decision Making Support for Parents and Caregivers

IRB Number Pro00111995

CRU/Department/Division/Center Department of Pediatrics

**Investigators** Monica Lemmon

Biostatistician(s) Analysis Biostatistician – Angel Davalos

Supervising Biostatistician – Hwanhee Hong

# 1. Study Overview

## **Background/Introduction**

The study is a single arm intervention trial for assessing the feasibility and acceptability a decision guide for parents of critically ill infants.

### Study Objectives, Aims, and Hypotheses

| Primary/ | Aim/Objective | Hypothesis |
|---|---|---|
| Secondary | | |
| Outcomes | | |
| Primary | Compute enrollment rate. | We expect the proportion of enrolled infants to |
| | | be at least 50%. |
| Primary | Compute complete data collection | We expect the proportion of enrolled families |
| | rate. | with data collected to be at least 80%. |
| Secondary | Describe decision aid | Descriptive objective, no hypothesis testing |
| | acceptability, stratified by parent | |
| | and clinician. | |
| Secondary | Describe pre- and post- parent | Descriptive objective, no hypothesis testing |
| | psychological distress, stratified by | |
| | parent. | |
| Secondary | Describe pre- and post- decision | Descriptive objective, no hypothesis testing |
| | (as appropriate) outcomes, | |
| | stratified by parent. | |
| Sample | Describe infant characteristics, | Descriptive objective, no hypothesis testing |
| description | parent demographics, and clinician | |
| | demographics. | |

# 2. Study Population and Data Source

#### **Study Design**

- Single arm design, study team will deliver a tool to be used by parent(s) to help guide them in decision making
- Tool includes a brief introduction to the tool and decision-making, a values clarification exercise, and a question prompt list
- Study will include: critically ill infants, their parent(s), and clinicians

#### **Inclusion Criteria**

- Infant inclusion criteria will include
  - 1. Age < 1 year
  - 2. Admission to a critical care unit
  - 3. Anticipated major decision

#### **Exclusion Criteria**

• Parent exclusion criteria will include 1) age < 18 years, 2) hearing or speech impairment, and 3) non-English speakers.

## **Data Acquisition**

• Data source: REDCap

• REDCap project name and ID: Decision Making PID 14854

# 3. Outcomes, Exposures, and Additional Variables of Interest

#### **Outcomes**

| Outcome | <b>Definition/Descriptions</b> | Variables and Source |
|---|---|---|
| Enrollment rate | Percentage of eligible infants enrolled. | screening log |
| Complete data collection rate | Complete data collection defined as all eligible infant, parent, and clinician data points collected for a given case; data points for which the participant withdrew prior to relevant data collection excluded | data collection log |
| PrepDM score | The preparation for decision making (PrepDM) scale evaluates parents' perceptions of how useful the decision aid was in preparing them to communicate with their child's health care team and make a decision. The 10-item survey uses a 5-point Likert scale. In accordance with the user manual and other studies, we will convert item responses to integers from 1 to 5, calculate the average, subtract 1 from average, and multiply by 25 to give a final score from 0 to 100. Higher scores indicate a higher perceived level of preparation for decision making. | prepdm_score (to be derived) Components: decision_present, decision_prep, consider_pros_cons, importance_pros_cons, depends_values, organize_thoughts, decision_involvement, questions_to_ask, discuss_values, prep_future_convos |

| Found this decision guide to be helpful | | guide_helpful |
|---|---|---|
| would recommend this decision guide to other parents making decisions about their child's health care | | rec_to_parents |
| would use this decision guide again if I need to make future decisions about my child's health care | | would_use_again |
| Promis t-score | We will measure scores for the following PROMIS domains: Short Form v2.0 Physical Function 4a, Short Form v1.0 Emotional Distress - Anxiety 8a, Short Form v1.0 Emotional Distress - Depression 8a, Short Form v1.0 Fatigue 4a, Short Form v1.0 Sleep Disturbance 4a, Short Form v2.0 Ability to Participate in Social Roles and Activities 4a, Short Form v1.1 Pain Interference 4a, and Numeric Rating Scale Pain Intensity 1a. The default calibration sample will be used for all scores. | stress_promis_tscore<br>(to be derived) |
| Family satisfaction in the intensive care unit (FS-ICU) | The decision making subscale of the FS-ICU is a 10-item survey that measures family surrogates' satisfaction with the decision making process in the ICU using 5-point Likert-type response formats. Families are asked to rate their satisfaction with communication from the health care team, the quality of the information they received, and how included and supported they felt in making medical decisions. In accordance with the survey's user manual and other studies, we will convert all item responses to integers from 0 to 4, calculate the average, and multiply by 25 to give a final score from 0 to 100. Aligning with prior studies from our group and others, a subscale score ≥75 will indicate a high level of satisfaction with decision making. | fs_icu (to be derived) |

| D | THE DDG: 61 | 1 (, 1 |
|---|---|---|
| Decisional regret score | The DRS is a 5-item survey that measures remorse or distress following a health care decision. Parents are asked to rate their agreement level with statements that express the presence or absence of regret, with 5 response options ranging from "strongly agree" to "strongly disagree." In accordance with the survey's user manual and other studies, we will convert all item responses to integers from 0 to 4, calculate the average, and multiply by 25 to give a final score from 0 to 100. Aligning with prior studies from our group and others, a score >25 will indicate a high level of decisional regret. | drs_score (to be derived) Components: drs_decisions, drs_regret, drs_again, drs_harm, drs_wise |
| Decisional conflict score | The DCS is a 16-item survey that measures parents' state of uncertainty about making health care decisions. Parents are asked to rate their agreement level with statements that relate to 5 domains of decisional conflict: being informed, support, effective decision making, uncertainty, and values clarity. In accordance with the survey's user manual and other studies, we will convert all item responses to integers from 0 to 4, calculate the average, and multiply by 25 to give a final score from 0 to 100. Aligning with prior studies from our group and others, a score >25 will indicate a high level of decisional conflict. | dcs_score (to be derived) Components: hard_v2, unsure_v2, clear_v2, awarechoice_v2, benefits_v2, risks_v2, advice_v2, importbene_v2, importrisk_v2, riskbenefit_v2, pressure_v2, amount_v2, informed_v2, selfdecision_v2, stick_v2, satisfied_v2 |
| Feeling heard<br>and understood<br>(FHAU) score | The 4-item FHAU scale measures parents' experience of feeling heard and understood by their infant's health care team using 5-point Likert-type response formats. In accordance with the user manual and other studies, we will use "top box scoring" for each item that defines "completely true" (i.e., the top box response) as passing, where 1 = passing and 0 = not passing. For each individual, we will average the number of top-box responses (up to 4) to estimate their proportion of Feeling Heard and Understood. We will also use descriptive statistics to calculate the total number of participants who responded "completely true" or "very true" for each item. | fhu_score (to be derived) Components: heard_understood, interests_first, interests_first, understood_values |

# 4. Statistical Analysis Plan

#### **Feasibility**

The primary outcome will be intervention and study feasibility, defined *a priori* as 1) enrollment rate of  $\geq 50\%$  of eligible infants and 2) complete data collection rate of  $\geq 80\%$ .

Enrollment rate will be computed as the number of infants enrolled divided by the number of eligible infants screened. Complete data collection will be defined as all eligible infant, parent, and clinician data points collected for a given case; data points for which a participant withdraws prior to relevant data collection will be excluded.

## Decision aid acceptability, Psychological stress, and Decision outcomes

Secondary outcomes include 1) parent and clinician acceptability of the tool, 2) preparation for decision-making, as measured by the Preparedness for Decision-making Scale (PrepDM), and 3) parent psychological distress, as measured using the PROMIS. Parent and clinician acceptability will be measured using self-report questions. Additional measured outcomes include parent decisional conflict, regret, and satisfaction. Decisional conflict and regret will be measured by the Decisional Conflict Scale (DCS) and the Decisional Regret Scale (DRS). Satisfaction with decision-making was measured using the Family Satisfaction-ICU decision-making subscale.

Decision aid acceptability will be summarized separately by parent, mother and father, as well as clinician. Pre- and post-intervention parental psychological stress and decision outcomes will be described for self-identified mothers and fathers separately.

Categorical characteristics will be summarized as frequency and percent, continuous characteristics will be summarized as mean, standard deviation, median, Q1, Q3, and range. A list of all reported variables can be found in the table shells in **section 5.** 

# 5. Appendix. Planned table shells:

| Table 1. Infant Characteristics | |
|---------------------------------|-------------------------|
| Characteristic | Median (Range) or n (%) |
| Infants enrolled (n=) | |
| Gestational age at birth, weeks | |
| Age at enrollment, days | |
| Sex, Female | |
| Medical condition | |
| Prematurity (<37 weeks) | |
| Seizures | |
| Genetic diagnosis | |
| Congenital heart disease | |
| Neurologic diagnosis | |
| Interventions (%) | |
| Mechanical ventilation | |
| Surgical feeding tube placement | |
| Palliative care consult | |
| Tracheostomy placement | |
| Length of hospital stay, days | |
| Location at enrollment | |
| NICU | |
| PCICU | |
| PICU | |
| Death during study enrollment | |

| <b>Table 2. Parent Characteristics</b> | |
|----------------------------------------|-------------------------|
| Characteristic | Median (Range) or n (%) |
| Parents enrolled (n=) | |
| Age, y | |
| Gender, Female | |
| Race and ethnicity | |
| African American | |
| Asian | |
| Hispanic/Latinx | |
| White | |
| More than one race | |
| Other/not reported | |
| Level of education | |
| Less than high school | |
| High school/GED | |
| Some college | |
| Bachelor's degree | |
| Associate's degree | |
| Graduate or professional degree | |
| Annual household income | |
| Less than \$25,000 | |
| \$25,000-\$34,999 | |
| \$35,000-\$49,999 | |
| \$50,000-\$74,999 | |
| \$75,000-\$99,999 | |
| \$100,000-\$149,999 | |
| Greater than \$150,000 | |
| Not reported | |
| Decision Guide Use | |
| Shared with clinical team | |
| Used in family conference | |

| Table 3. Clinician Characteristics | |
|------------------------------------|-------------------------|
| Characteristic | Median (Range) or n (%) |
| Clinicians enrolled (n=) | |
| Age, y | |
| Gender, Female | |
| Race and ethnicity | |
| African American | |
| Asian | |
| Hispanic/Latinx | |
| White | |
| More than one race | |
| Other/not reported | |
| Years in practice | |
| Specialty | |
| Neonatology | |
| Pediatric critical care | |
| Pediatric neurology | |
| Pediatric cardiology | |
| Neurosurgery | |
| Other | |
| Social work | |
| Nursing | |
| Decision Guide Acceptability | |
| Found it to be helpful | |
| Would recommend to parents | |
| Would use again in future | |

| Table 4. Decision Aid Acceptability | | | |
|---|---|---|---|
| Acceptability measure | Mothers | Fathers | Clinicians |
| Found to be helpful | | | |
| Would recommend to other parents/patients | | | |
| Would use in the future | | | |

Categorical variables display n for Agree/Strongly agree.

| Table 5. Preparedness for Decision Making | | | |
|---|---|---|---|
| | Mothers | Fathers | Clinicians |
| PrepDM score | | | |
| PrepDM items (n agree or strongly agree, %) | | | |
| Helped recognize that decision needs | | | |
| to be made for child | | | |
| Prepared me to make decision for child | | | |
| Helped me think about the pros and | | | |
| cons of each treatment option | | | |
| Helped me think about which pros and | | | |
| cons are most important | | | |
| Helped me know that the decision | | | |
| depends on what matters most to me | | | |
| Helped me organize my thoughts | | | |
| Helped me think about how involved I | | | |
| want to be in making decisions | | | |
| Helped me identify questions to ask | | | |
| my child's doctor | | | |
| Prepared me to talk to my child's | | | |
| doctor about what matters most to me | | | |
| Prepared me for future conversations | | | |
| with my child's doctor | | 3.4 : 1 | |

Median (IQR) and n (%) for continuous and categorical variables, respectively. Categorical variables display n for Agree/Strongly agree or Quite a bit/A great deal

| Table 6. Parent well-being (PROMIS measure) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline | Baseline | | | Post-Intervention | | | Difference (Post - Pre) | |
| Score | Response | Baseline<br>Mother | Baseline<br>Father | Baseline All<br>Participants | Post-<br>Intervention<br>Mother | Post-<br>Intervention<br>Father | Post-<br>Intervention<br>All<br>Participants | Post - Pre<br>Mother | Post - Pre<br>Father | Post - Pre<br>All<br>Participants |
| PROMIS: Ability to Participate in Social Roles and Activities | | | | | | | | | | |
| PROMIS: Emotional Distress –<br>Anxiety | | | | | | | | | | |
| PROMIS: Emotional Distress –<br>Depression | | | | | | | | | | |
| PROMIS: Fatigue | | | | | | | | | | |
| PROMIS: Pain Intensity | | | | | | | | | | |
| PROMIS: Pain Interference | | | | | | | | | | |
| PROMIS: Physical Function | | | | | | | | | | |

Median (IQR) and n (%) for continuous and categorical variables, respectively.

PROMIS: Sleep Disturbance

| Table 7. Decisional conflict, decisional regret, decision-making satisfaction, and feeling heard and understood. | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline | | | Post-Intervention | | | Difference (Post - Pre) | | |
| Score | Response | Baseline<br>Mother | Baseline<br>Father | Baseline All<br>Participants | Post-<br>Intervention<br>Mother | Post-<br>Intervention<br>Father | Post-<br>Intervention<br>All<br>Participants | Post - Pre<br>Mother | Post - Pre<br>Father | Post - Pre<br>All<br>Participants |
| Decisional Conflict score | | | | | | | | | | |
| Effective Decision | | | | | | | | | | |
| Informed | | | | | | | | | | |
| Support | | | | | | | | | | |
| Uncertainty | | | | | | | | | | |
| Values Clarity | | | | | | | | | | |
| Decisional Regret score | | | | | | | | | | |
| Family Satisfaction-ICU score | | | | | | | | | | |
| Feeling Heard and Understood score | | | | | | | | | | |

Median (IQR) and n (%) for continuous and categorical variables, respectively. Categorical variables display n for Agree/Strongly agree or Quite a bit/A great deal.